CLINICAL TRIAL: NCT05687435
Title: Changyanning Tablet for the Treatment of Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D): A Multicenter, Randomized, Double Blind, Placebo-Controlled Trial
Brief Title: Changyanning Tablet for the Treatment of Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mei Han (Other)
Responsible Party: Sponsor-Investigator, Mei Han, Principal Investigator, Beijing University of Chinese Medicine
Organization: Beijing University of Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CYNT-2022-12
Record Dates: First submitted 2022-12-23; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Diarrhea-Predominant Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Changyanning group (Experimental): Changyanning tablet: Each tablet weighs 0.42g and is taken orally, 4 tablets once and 3 times a day.The course of treatment was 8 weeks.
  Interventions: Drug: Changyanning tablet
- Placebo group (Placebo Comparator): Changyanning tablet placebo: Each tablet weighs 0.42g and is taken orally, 4 tablets once and 3 times a day.The course of treatment was 8 weeks.
  Interventions: Other: Changyanning tablet placebo

INTERVENTIONS:
Drug: Changyanning tablet — Changyanning Tablet is produced by Jiangxi Kang'enbei Traditional Chinese Medicine Co., Ltd，composed of Euphorbia humifusa, golden ear grass, camphor tree root, Elsholtzia splendens and maple leaves. It is mainly used for the treatment of acute and chronic intestinal diseases caused by various reasons.
  If the symptoms of the subject become worse and unbearable during the study period, it is allowed to add Pinaverium Bromide to the patient according to the specific situation.
  Arms: Changyanning group
Other: Changyanning tablet placebo — Changyanning Tablet placebo is produced by Jiangxi Kang'enbei Traditional Chinese Medicine Co., Ltd. Changyanning Tablet placebo has the same appearance, smell, taste, specifications and packaging with Changyanning Tablet, but does not contain active pharmaceutical ingredients.
  If the symptoms of the subject become worse and unbearable during the study period, it is allowed to add Pinaverium Bromide to the patient according to the specific situation.
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to test the efficacy and safety of the Chinese patent medicine Changyanning Tablet in the patients with Diarrhea-Predominant Irritable Bowel Syndrome (IBS-D). The main questions it aims to answer are:

1. Can Changyanning Tablet improve diarrhea and abdominal pain in IBS-D patients?
2. Is Changchangning Tablet safe for the treatment of IBS-D?

ELIGIBILITY:
Inclusion Criteria:

1. Meet IBS-D Rome IV diagnostic criteria;
2. Age between 18 and 65 years old (including boundary value), regardless of gender;
3. IBS symptom severity scale (IBS-SSS) scores > 175 points;
4. The weekly average score of abdominal pain in screening period is ≥ 3 points (The most severe abdominal pain in the past 24 hours every day, the pain score was 11 grades (0-10), NRS-11; Also the number of days of the stool character classification (Bristol stool scale) is type 6 or 7 ≥ 2 in a week;
5. Patients who voluntarily accept the program's plan of the project and signs the informed consent form.

Exclusion Criteria:

1. Patients with serious or unstable heart, liver, kidney, immune, endocrine system and other diseases or malignant tumors;
2. Patients are affected by factors such as intellectual disorder, mental disorder and language;
3. Patients with gastrointestinal organic diseases or with malignant tumors, such as pancreatitis, intestinal adenoma (excluding polypectomy for more than half a month), intestinal diverticulum, colon or rectal cancer, inflammatory bowel disease, intestinal tuberculosis, etc;
4. Other diseases (such as hyperthyroidism, diabetes, chronic renal insufficiency, nervous system diseases, etc.) that affect digestive tract dynamics;
5. Complicated with tuberculosis peritonitis, gallstones, cirrhosis, chronic pancreatitis and other gastrointestinal diseases;
6. Allergic constitution or allergic to the components of the studied drug;
7. Pregnant or lactating women, and women with recent fertility plans;
8. Previous abdominal or pelvic surgery, such as cholecystectomy;
9. Patients with positive fecal occult blood;
10. During the screening period, drugs that affect gastrointestinal motility and function cannot be stopped, including parasympathetic inhibitors, such as scopolamine, atropine, belladonna, etc; Muscle relaxants, such as succinylcholine; Antidiarrheal agents such as loperamide, smecta, etc; Opioid preparations, etc;
11. Those who use probiotics (except those who eat yoghurt) or antibiotics within 8 weeks before enrollment in the study;
12. IBS drugs (except polyethylene glycol and loperamide) were used within 3 months before the study;
13. Those who regularly drink alcohol within 6 months before screening, i.e., drink more than 14 units of alcohol every week (1 unit=360 mL beer or 45 mL liquor or 150 mL wine with 40% alcohol);
14. Those who have participated in or are currently participating in other clinical trials within 1 month before screening;
15. The researcher believes that there are patients who are not suitable for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-01-30 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Weekly response rate of abdominal pain and diarrhea | 8 weeks (after treatment)
  The responder is defined when the following two points are met simultaneously： ① Abdominal pain intensity: the most severe abdominal pain score in the past 24 hours, the weekly average value is at least 30% lower than the baseline. To evaluate the intensity of abdominal pain, the patients were asked to grade "the most severe abdominal pain in the past 24 hours" every day by using the 0-10 numerical rating scale (NRS).
  ② Fecal traits: the number of days with type 6 or 7 stool traits in a week decreased by at least 50% from the baseline. Refer to Bristol Stool Traits Scale for evaluation of fecal traits.
  The response rate=(the number of the responders/the sample size of the group) x100%.

SECONDARY OUTCOMES:
Weekly response rate of abdominal pain and diarrhea | 2 weeks, 4 weeks, 6 weeks, 12 weeks
  The responder is defined when the following two points are met simultaneously： ① Abdominal pain intensity: the most severe abdominal pain score in the past 24 hours, the weekly average value is at least 30% lower than the baseline. To evaluate the intensity of abdominal pain, the patients were asked to grade "the most severe abdominal pain in the past 24 hours" every day by using the 0-10 numerical rating scale (NRS).
  ② Fecal traits: the number of days with type 6 or 7 stool traits in a week decreased by at least 50% from the baseline. Refer to Bristol Stool Traits Scale for evaluation of fecal traits.
  The response rate=(the number of the responders/the sample size of the group) x100%.
Weekly response rate of diarrhea | 2 weeks, 4 weeks, 6 weeks, 8 weeks，12 weeks
  The responder is defined when the following two points are met simultaneously： ①Fecal traits: the number of days with type 6 or 7 stool traits in a week decreased by at least 50% from the baseline. Refer to Bristol Stool Traits Scale for evaluation of fecal traits.
  ②Abdominal pain intensity: the most severe abdominal pain score in the past 24 hours, the weekly average value is remained unchanged or improved from baseline. To evaluate the intensity of abdominal pain, the patients were asked to grade "the most severe abdominal pain in the past 24 hours" every day by using the 0-10 numerical rating scale (NRS).
  The response rate=(the number of the responders/the sample size of the group) x100%.
Weekly response rate of abdominal pain | 2 weeks, 4 weeks, 6 weeks, 8 weeks，12 weeks
  The responder is defined when the following two points are met simultaneously： ①Abdominal pain intensity: the most severe abdominal pain score in the past 24 hours, the weekly average value is at least 30% lower than the baseline. To evaluate the intensity of abdominal pain, the patients were asked to grade "the most severe abdominal pain in the past 24 hours" every day by using the 0-10 numerical rating scale (NRS).
  ②Fecal traits: the number of days and frequency with type 6 or 7 stool traits in a week is remained unchanged or decreased from baseline. Refer to Bristol Stool Traits Scale for evaluation of fecal traits.
  The response rate=(the number of the responders/the sample size of the group) x100%.
IBS symptom severity scale（IBS-SSS）scores | 2 weeks, 4 weeks, 6 weeks, 8 weeks，12 weeks
  There are five questions in the scale, each of which has a full score of 100 points and a total score of 500 points. The higher the total score, the more serious the patient's symptoms.
Stool frequency | 2 weeks, 4 weeks, 6 weeks, 8 weeks，12 weeks
  Daily average number of spontaneous defecation in a week.
IBS quality of life (IBS-QOL) scores | 6 weeks, 8 weeks（after treatment），12 weeks（after follow-up）
  The scale consists of 34 items, and each item is divided into five grades: asymptomatic, mild, moderate, overweight, and severe, with corresponding scores of 1-5. The higher the total score, the more serious the patient's symptoms.

OTHER OUTCOMES:
Blood routine test | baseline， 8weeks（after treatment）
  This is a safety outcome.
C-reactive protein | baseline， 8weeks（after treatment）
  This is a safety outcome.
Urine routine test | baseline， 8weeks（after treatment）
  This is a safety outcome.
Stool routine test | baseline， 8weeks（after treatment）
  This is a safety outcome.
Stool occult blood | baseline， 8weeks（after treatment）
  This is a safety outcome.
Liver function-Alanine aminotransferase（ALT） | baseline， 8weeks（after treatment）
  This is a safety outcome.
Liver function-Aspartate aminotransferase (AST) | baseline， 8weeks（after treatment）
  This is a safety outcome.
Liver function-alkaline phosphatase (ALP) | baseline， 8weeks（after treatment）
  This is a safety outcome.
Renal function-blood urea nitrogen (BUN) | baseline， 8weeks（after treatment）
  This is a safety outcome.
Renal function-creatinine | baseline， 8weeks（after treatment）
  This is a safety outcome.
Electrocardiogram | baseline， 8weeks（after treatment）
  This is a safety outcome.
Adverse events | Up to 8 weeks
  This is a safety outcome.
Serious adverse events | Up to 8 weeks
  This is a safety outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wei, Pro, Principal Investigator — Wangjing Hospital of China Academy of Chinese Medical Sciences

IPD SHARING:
Plan to Share IPD: No